CLINICAL TRIAL: NCT06731530
Title: A Comparative Study of Anterior Segment Structural Features, Biomechanical Behaviour and Optical Properties of the Cornea in Patients With and Without Pseudoexfoliation Syndrome.
Brief Title: Corneal Biomechanics, Optical Properties and Anterior Segment Structural Features in Patients With Pseudoexfoliation
Acronym: CorPEX
Status: Recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Papageorgiou General Hospital (Other)
Responsible Party: Principal Investigator, Nikolaos Ziakas, Professor of Ophthalmology, Aristotle University Of Thessaloniki
Other Study IDs: 36661
Record Dates: First submitted 2024-11-19; First posted 2024-12-12 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pseudoexfoliation Syndrome; Biomechanical Parameters; Corneal Densitometry
Keywords: pseudoexfoliation syndrome; biomechanical parameters; corneal transparency
MeSH Terms: conditions — Exfoliation Syndrome | interventions — Slit Lamp

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PEX group (patients WITH pseudoexfoliation syndrome): right or left eye of pseudophakic patients diagnosted with PEX syndrome pre-operatively (PEX positive, as recorded in the pre-operative medical file)
  Interventions: Device: Pentacam-AXL; Device: HD Analyzer; Device: Corvis ST; Device: OCT-A Angiovue; Device: IOLMaster V.5.4; Device: Topcon SP-1P; Other: BCVA (ETDRS), Slit lamp examination, Goldmann Applanation Tonometry, Fundus examination
- Control group (patients WITHOUT pseudoexfoliation syndrome): right or left eye of pseudophakic patients without a pre-operative diagnosis of pseudoexfoliation syndrome (PEX negative, as recorded in the pre-operative medical file)
  Interventions: Device: Pentacam-AXL; Device: HD Analyzer; Device: Corvis ST; Device: OCT-A Angiovue; Device: IOLMaster V.5.4; Device: Topcon SP-1P; Other: BCVA (ETDRS), Slit lamp examination, Goldmann Applanation Tonometry, Fundus examination

INTERVENTIONS:
Device: Pentacam-AXL — Pentacam-AXL (Oculus, Wetzlar, Germany)
Device: HD Analyzer — HD Analyzer (Visiometrics, Terassa, Spain, Keeler)
Device: Corvis ST — Corvis ST (Oculus, Germany)
Device: OCT-A Angiovue — OCT-A Angiovue (Optovue, Inc., Fremont, California, USA)
Device: IOLMaster V.5.4 — IOLMaster V.5.4 (Carl Zeiss., Meditec)
Device: Topcon SP-1P — Topcon SP-1P (Topcon Medical Inc., Tokyo, Japan)
Other: BCVA (ETDRS), Slit lamp examination, Goldmann Applanation Tonometry, Fundus examination — BCVA (ETDRS), Slit lamp examination, Goldmann Applanation Tonometry, Fundus Examination

SUMMARY:
The purpose of this study is to assess the effect of pseudoexfoliation syndrome on corneal biomechanics, optical clarity of the cornea, and anterior segment structural features.

DETAILED DESCRIPTION:
A case group of patients with pseudoexfoliation syndrome will ungergo examinations to evaluate corneal optical properties (Pentacam-AXL, HD analyzer), biomechanics (Corvis ST) and anterior segment structural features (OCT-A Angiovue, Pentacam-AXL, IOLMaster V.5.4, Topcon SP-1P). The same examinations will be performed on a group of age-matched controls, and the results will be compared.

Corneal optical density will be assessed by backscatter measurement (COD, corneal optical density) using Pentacam AXL (Oculus, Wetzlar, Germany).

Corneal optical density will also be assessed by forward-scatter measurement (OSI, objective scatter index) using HD Analyzer (Visiometrics, Terassa, Spain, Keeler). The level of agreement between the two optical density indicators (OSI, COD) will be evaluated.

Corneal biomechanics measurements will be performed using Corvis Scheimpflug Technology. The main biomechanical parameter of the Corvis ST is DA (deformation amplitude). DA quantifies how the cornea deforms in response to an air puff and helps evaluate corneal stiffness and elasticity.

An additional objective is the study of structural parameters of the cornea as well as, more broadly, the anterior segment in pseudoexfoliation syndrome (PEX) patients, aiming to understand and describe the effects of PEX with the highest possible accuracy. Specifically, using the Pentacam-AXL (Oculus, Wetzlar, Germany), the IOLMaster V.5.4 (Carl Zeiss Meditec), the OCT-Angiography Angiovue (Optovue, Inc., Fremont, California, USA), and the specular microscope Topcon SP-1P (Topcon Medical Inc., Tokyo, Japan), a comparative study will be conducted across a range of variables and maps: corneal topographic data, keratometric measurements, curvature radius data, pachymetric data, anterior chamber depth and volume, angle width, axial length, pupil diameter, and endothelial cell density. Some of these data, such as central corneal thickness, can be measured by two of the aforementioned devices. In this case, we will also attempt to evaluate the level of agreement between the two devices.

ELIGIBILITY:
Inclusion Criteria:

* age 60-80 years.
* unilateral or bilateral pseudophakia (cataract surgery undergone at Papageorgiou General Hospital, Thessaloniki, Greece).
* open anterior chamber angle (grade > 2, van Herick method).

Exclusion Criteria:

* History of intraocular surgery other than uncomplicated cataract surgery (phakoemulsification).
* Cataract surgery within the last 3 months.
* History of ocular trauma.
* Use of contact lenses.
* Corneal pathology.
* Use of anti-VEGF medications.
* History of uveitis or active uveitis.
* Hypertension (IOP > 21 mmHg) or glaucoma.
* Myopia or hyperopia greater than 3 diopters.
* Astigmatism greater than 1.5 diopters.
* Posterior capsular opacification grade 2, 3, or 4 based on the EPCO grading scale.
* Tear break-up time <10 sec

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from patients who consult at the outpatient clinic of the 2nd Department of Ophthalmology, General Hospital Papageorgiou, Thessaloniki, Greece.
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Corneal optical density assessed by backscatter measurement | Baseline, during examination : approx. 1 hour
  Corneal optical density assessed by backscatter measurement (COD, corneal optical density) using Pentacam AXL (Oculus, Wetzlar, Germany)
Corneal optical density assessed by forward-scatter measurement | Baseline, during examination : approx. 1 hour
  Corneal optical density assessed by forward-scatter measurement (OSI, objective scatter index) using HD Analyzer (Visiometrics, Terassa, Spain, Keeler)

SECONDARY OUTCOMES:
Corneal biomechanics using Corvis Scheimpflug Technology | Baseline, during examination : approx. 1 hour
  The main biomechanical parameter of the Corvis ST : DA (deformation amplitude). DA quantifies how the cornea deforms in response to an air puff and helps evaluate corneal stiffness and elasticity.
Optical quality measured by HD-analyzer : Strehl ratio | Baseline, during examination : approx. 1 hour
  Specific measurement variable: Total score of Strehl ratio; Value [no dimension];
Optical quality measured by HD-analyzer : MTF cut-off | Baseline, during examination : approx. 1 hour
  Specific measurement variable: Total score of Modulation transfer function (MTF) cut-off; Value [c/deg];
Corneal biomechanics using Corvis Scheimpflug Technology : velocity | Baseline, during examination : approx. 1 hour
  Velocity during the first and the second applanation of the cornea, measured using Corvis ST [m/s]
Corneal biomechanics using Corvis Scheimpflug Technology : length | Baseline, during examination : approx. 1 hour
  First and second applanation length (mm)
Corneal biomechanics using Corvis Scheimpflug Technology : bIOP | Baseline, during examination : approx. 1 hour
  Biomechanically corrected IOP (bIOP) (mmHg)

OTHER OUTCOMES:
The level of agreement between the two optical density indicators (OSI, COD) after standardization | Baseline, during examination : approx. 1 hour
  The level of agreement between the two optical density indicators : objective scatter index (OSI), corneal optical density (COD) after standardization. Value [no dimension]
Anterior chamber depth (mm) | Baseline, during examination : approx. 1 hour
  Anterior chamber depth (mm)
Endothelial cell density (cells/mm2) | Baseline, during examination : approx. 1 hour
  Endothelial cell density (cells/mm2)
Corneal topography (D) | Baseline, during examination : approx. 1 hour
  Corneal topography (D)
Anterior chamber volume (mm3) | Baseline, during examination : approx. 1 hour
  Anterior chamber volume (mm3)
Anterior chamber angle (°) | Baseline, during examination : approx. 1 hour
  Anterior chamber angle (°)
Axial length (mm) | Baseline, during examination : approx. 1 hour
  Axial length (mm)
Central corneal thickness (μm) | Baseline, during examination : approx. 1 hour
  Central corneal thickness (μm)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Ziakas, Professor, Study Chair — Aristotle University Of Thessaloniki
Locations (1):
- 2nd Department of Ophthalmology, Papageorgiou General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
Deidentified Individual Participant Data (IPD) that underline published results, along with related data dictionaries, will be available only to researchers who will provide a methodologically sound proposal, after acceptance of the proposed protocol by our Institution's IRB. Data requestors will need to sign a data access agreement. The study protocol and statistical analysis plan will also be available, if needed.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months.
Access Criteria: Available only to researchers who will provide a methodologically sound proposal, after acceptance of the proposed protocol by our Institution's IRB. Data requestors will need to sign a data access agreement.